CLINICAL TRIAL: NCT06531603
Title: Comparison of Postoperative Analgesic Effectiveness of Bupivacaine and Bupivacaine Plus Dexmedetomidine Wound Infiltration in Abdominal Surgeries Under General Anesthesia
Brief Title: Postoperative Analgesic Effectiveness of Bupivacaine With and Without Dexmedetomidine in Patients With Abdominal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Principal Investigator, Muhammad Shahid, Associate Professor, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB29
Record Dates: First submitted 2024-07-03; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain; Bradycardia; Hypotension; Nausea; Vomiting
Keywords: Bupivacaine; Dexmedetomidine; Post operative analgesia; Abdominal surgery
MeSH Terms: conditions — Pain, Postoperative; Bradycardia; Hypotension; Nausea; Vomiting | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and assessor were unaware of interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine group (Experimental): Patients receiving Bupivacaine plus placebo for wound infiltration after abdominal surgery for pain control.
  Interventions: Drug: bupivacaine wound infilteration
- Bupivacaine plus Dexmedetomidine group (Experimental): Patients receiving Bupivacaine plus Dexmedetomidine for wound infiltration after abdominal surgery for pain control.
  Interventions: Drug: Bupivacaine plus dexmedetomidine wound infilteration

INTERVENTIONS:
Drug: bupivacaine wound infilteration — drug was given at the end of surgery
  Other Names: LA infiltration
  Arms: Bupivacaine group
Drug: Bupivacaine plus dexmedetomidine wound infilteration — drug was given at the end of surgery
  Other Names: LA + Dex infiltration
  Arms: Bupivacaine plus Dexmedetomidine group

SUMMARY:
Abdominal surgeries are major surgical procedures that are performed at any teaching hospital. Pain control is major concern in the intra-operative as well as post-operative period in these patients. Optimal pain control in post-operative period is directly related to patient's recovery, shortens the patients' hospital stay and overall burden on health facilities. Inadequate pain control may affect quality of life and increases patient's morbidity and mortality. Different modalities for pain control are used in post-operative period. Opioids are mainstay of treatment in post-operative period but historically are associated with significant side effect profile like dependence, nausea, vomiting, respiratory depression, constipation and many others. Dexmedetomidine is centrally acting α-2 adrenoceptor agonist.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted at Department of Anesthesia, Sahiwal Teaching Hospital, Sahiwal. After institutional review board (IRB) approval, computer-generated random number table was used to randomize the patients to two groups, one group received Bupivacaine plus placebo and the other group received Bupivacaine plus dexmedetomidine. A total of 64 patients met the inclusion criteria and were enrolled in the study in a 1:1. Informed written consent was obtained from all the patients before enrolling them in the study. All patients underwent a pre-operative assessment on the day before surgery. Both groups received wound infiltration with studied drugs at the end of surgery. After surgery patients were shifted to post-surgical ward and assessed for pain using visual analogue scale (VAS) and data was collected and analyzed using Statistical Package for the Social Sciences (SPSS) version 26. Quantitative variables were presented with mean ±SD. Comparison of quantitative variable between groups was done using independent sample t-test. Comparison of qualitative variable like (Opioid sparing effect, Bradycardia, Hypotension, Nausea, Vomiting) was presented with frequency and percentages. Data was stratified on the basis of gender and age. Post-stratification chi-square test was used to compare both groups for opioid sparing effect in each stratum with p-value ≤0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age limit: 18-60 years
2. Gender of patient i.e., male or female
3. Patients listed for abdominal surgeries
4. American Society of Anesthesiologists (ASA) status of I or II

Exclusion Criteria:

1. Patients with history of drug allergy
2. Patients who undergone any analgesia in past 24 hr
3. Patients with liver disease, kidney disease, cardiac disease, sickle cell anemia, severe preeclampsia or CNS disorder on history, clinical and laboratory assessment
4. American Society of Anesthesiologists (ASA) status III or IV
5. Patients with morbid obesity 6, Raynaud's disease Patients on adrenoceptor agonists, antagonists or narcotics before the operation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | Every 30 mints for 4hrs than 2hrly for 24 hrs post procedure
  Time from procedure to requirement of rescue analgesia

SECONDARY OUTCOMES:
Opioid sparing | Total dose of nalbuhine consumption in 1st 24 hrs after procedure
  Total amount of opioid consumtion in the first 24 post procedure.
Blood pressure | Every 15 minutes intra operative and every 15 minutes for 24 hrs postoperatively
  Mean pressue will be measured
Hear rate | Every 15 minutes intraoperative and every 15 minutes postoperatively for 24 hrs
  Heart rate will be measured
Neausea | Every 30 minutes for 4 hrs then 2hrly for 24 hrs
  Felling of nasueas
Vomiting | Every 3 minutes for first 4 hrs then 2hrly for 24 hrs
  Urge to vomit

CONTACTS AND LOCATIONS:
Overall Officials: M. Shahid, FCPS, Principal Investigator — Sahiwal medical college sahiwal; A. Riaz, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- Sahiwal Medical College, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
We will not share individualized data, but the outcomes of the study will be shared in the form of manuscript.

REFERENCES:
- [Result] Chen J, Zhou JQ, Chen ZF, Huang Y, Jiang H. Efficacy and safety of dexmedetomidine versus propofol for the sedation of tube-retention after oral maxillofacial surgery. J Oral Maxillofac Surg. 2014 Feb;72(2):285.e1-7. doi: 10.1016/j.joms.2013.10.006. Epub 2013 Oct 25. PMID 24438599
- [Result] Champaneria R, Shah L, Geoghegan J, Gupta JK, Daniels JP. Analgesic effectiveness of transversus abdominis plane blocks after hysterectomy: a meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2013 Jan;166(1):1-9. doi: 10.1016/j.ejogrb.2012.09.012. Epub 2012 Oct 4. PMID 23041302
- [Result] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Result] Brogi E, Kazan R, Cyr S, Giunta F, Hemmerling TM. Transversus abdominal plane block for postoperative analgesia: a systematic review and meta-analysis of randomized-controlled trials. Can J Anaesth. 2016 Oct;63(10):1184-1196. doi: 10.1007/s12630-016-0679-x. Epub 2016 Jun 15. PMID 27307177
- [Result] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Result] Bhatia N, Arora S, Jyotsna W, Kaur G. Comparison of posterior and subcostal approaches to ultrasound-guided transverse abdominis plane block for postoperative analgesia in laparoscopic cholecystectomy. J Clin Anesth. 2014 Jun;26(4):294-9. doi: 10.1016/j.jclinane.2013.11.023. Epub 2014 Jun 2. PMID 24882606
- [Result] Bhananker SM, Posner KL, Cheney FW, Caplan RA, Lee LA, Domino KB. Injury and liability associated with monitored anesthesia care: a closed claims analysis. Anesthesiology. 2006 Feb;104(2):228-34. doi: 10.1097/00000542-200602000-00005. PMID 16436839
- [Result] Ayad S, Babazade R, Elsharkawy H, Nadar V, Lokhande C, Makarova N, Khanna R, Sessler DI, Turan A. Comparison of Transversus Abdominis Plane Infiltration with Liposomal Bupivacaine versus Continuous Epidural Analgesia versus Intravenous Opioid Analgesia. PLoS One. 2016 Apr 15;11(4):e0153675. doi: 10.1371/journal.pone.0153675. eCollection 2016. PMID 27082959
- [Result] Ard JL Jr, Bekker AY, Doyle WK. Dexmedetomidine in awake craniotomy: a technical note. Surg Neurol. 2005 Feb;63(2):114-6; discussion 116-7. doi: 10.1016/j.surneu.2004.02.029. PMID 15680647
- [Result] Arain SR, Ebert TJ. The efficacy, side effects, and recovery characteristics of dexmedetomidine versus propofol when used for intraoperative sedation. Anesth Analg. 2002 Aug;95(2):461-6, table of contents. doi: 10.1097/00000539-200208000-00042. PMID 12145072
- [Result] Altuntas G, Akkaya OT, Ozkan D, Sayin MM, Balas S, Ozlu E. Comparison of Intraabdominal and Trocar Site Local Anaesthetic Infiltration on Postoperative Analgesia After Laparoscopic Cholecystectomy. Turk J Anaesthesiol Reanim. 2016 Dec;44(6):306-311. doi: 10.5152/TJAR.2016.75983. Epub 2016 Dec 1. PMID 28058142
- [Result] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518
- [Result] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424

DOCUMENTS (1):
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT06531603/ICF_000.pdf